CLINICAL TRIAL: NCT05176652
Title: Reliability of Utrasonographic Diameter of Optic Nerve Sheath in Assessment of Fluid Status in Severe Preeclamptic Patients
Brief Title: Ultrasonographic Diameter of Optic Nerve Sheath in Fluid Assessment in Severe Preeclamptic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hossam Eldin Hassan Ahmed, assisstant lecturer of anesthesia and ICU ,faculty of medicine at sohag university, Sohag University
Other Study IDs: Soh-Med-21-12-21
Record Dates: First submitted 2021-12-14; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Severe Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: ultrasound — ultrasonographic assessment of optic nerve sheath diameter

SUMMARY:
Changes in the optic nerve sheath diameter detected by ultrasound are considered an important manifestation of increased intracranial pressure . The normal optic nerve sheath diameter measures up to 5.0 mm and an average optic nerve sheath diameter more than 5 mm is considered abnormal and elevated intracranial pressure should be suspected.Cerebral edema have been demonstrated in 71% to 100% of magnetic resonance imaging in preeclamptic patients and an increase in optic nerve sheath diameter has been described in preeclamptic females compared to healthy pregnant females Therefore, Increased optic nerve sheath diameter can indirectly reflect the state of intracranial edema that could be a part of generalized edema of preeclampsia and it could be a possible marker of generalized tissue edema and fluid overload in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure of 160mm Hg or higher, or diastolic blood pressure of 110mm Hg or higher on 2 occasions at least 6 hours apart on bed rest.
* Proteinuria ≥5g in a 24 hour urine specimen or ≥3+ on 2 random urine samples collected at least 4 hours apart.
* patient acceptance
* Accepted mental state of the patients

Exclusion Criteria:

* patient refusal to participate in the study
* chronic kidney disease
* chronic pulmonary disease
* chronic cardiac disease
* chronic hypertension
* previous ocular operation and diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant preeclamptic patients
Study Population: severe preeclamptic patients (aged 18-40) after termination of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-10-06 (Estimated); Study Completion 2022-12-06 (Estimated)

PRIMARY OUTCOMES:
correlation between optic nerve sheath diameter and extravascular lung water | up to 24 hours
  correlation between ultrasound assessment of optic nerve sheath diameter and extravascular lung water

CONTACTS AND LOCATIONS:
Locations (1):
- Hossam Eldin Hassan Ahmed Abdelghani, Sohag, Egypt